CLINICAL TRIAL: NCT03179501
Title: Effect of Single Dose NP001 on Blood Markers of Inflammation in Individuals With Mild-to-Moderate Alzheimer's Disease
Brief Title: NP001, Alzheimer's Disease, and Blood Markers of Inflammation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Beau Nakamoto (Other)
Collaborators: Neuraltus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Beau Nakamoto, Associate Professor, Department of Medicine, John A. Burns School of Medicine, University of Hawaii at Manoa, University of Hawaii
Organization: University of Hawaii (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H039
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Single-site, randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NP001 (Experimental): NP001
  Interventions: Drug: NP001
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NP001 — NP001
  Arms: NP001
Drug: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
This is a Phase 1 placebo-controlled biomarker study of NP001 in individuals with Alzheimer's Disease.

DETAILED DESCRIPTION:
Abnormal inflammatory monocytes/macrophages, systemically and locally in the central nervous system (CNS), are implicated in the neuro-inflammatory process seen in Alzheimer's disease. NP001 is a novel immune regulator of inflammatory monocytes/macrophages.

Given the key role inflammatory monocytes/macrophages may play in the pathogenesis of AD, this study will assess the changes in inflammatory monocyte-associated biomarkers, including CD16 and HLA-DR, pre- and post- NP001.

This is a Phase 1 single-site, randomized, double-blind, placebo-controlled pilot biomarker study of a single dose of NP001 in individuals with mild-to-moderate Alzheimer's disease. Fourteen individuals will be enrolled and randomized 1:1 to NP001 and placebo. Drug or placebo will be given intravenously. Biomarkers will be measured at baseline and 1 and 7 days following infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 55 years of age or older,
2. Diagnosis of probable Alzheimer's disease using the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's disease and Related Disorders Association criteria by Principal Investigator,
3. Score 14 to 24 (inclusive) on the Mini-Mental Status Examination,
4. Global Clinical Dementia Rating (CDR) Scale ≥ 0.5 or greater with CDR memory ≥ 0.5 or greater,
5. Score ≤ 4 or lower on the Hachinski Ischemic Scale,
6. Score ≤ 5 on the Geriatric Depression Scale (GDS),
7. Current (stable dose for 4 weeks or longer) or past treatment with acetylcholinesterase inhibitors, memantine, or cognitive enhancers are allowed,
8. Females must not be of childbearing potential (i.e., must be post-menopausal with cessation of menses for ≥ 12 months or have been surgically sterilized which includes hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or tubal ligation),
9. Males must agree not to engage in sexual relations with a woman of childbearing potential without effective means of birth control during the study and for 30 days after study drug administration. Must also agree to refrain from sperm donation from receipt of study drug and for 90 days thereafter.
10. Be capable of providing written informed consent using a form that has been approved by the IRB.
11. Have veins suitable for intravenous administration of study drug or alternatively, have a venous access device.

Exclusion Criteria:

1. Diagnosis of another neurologic disorder which can mimic Alzheimer's disease including dementia with Lewy Bodies, frontotemporal dementia and normal pressure hydrocephalus,
2. Diagnosis of other neurologic disorders which can also impair cognition including stroke, MS, seizures, CNS tumors,
3. Uncontrolled major psychiatric disorder,
4. History of unstable medical illness in the 3 months prior to screening including emergent hospitalizations,
5. Diagnosis of any of the following disorders: systemic sclerosis/scleroderma, inflammatory bowel disease, systemic lupus erythematosus (SLE), rheumatoid arthritis, mixed connective tissue disease, polymyalgia rheumatica, giant cell arteritis, polymyositis, dermatomyositis, and psoriasis,
6. Active pulmonary disease under treatment including uncontrolled asthma, chronic obstructive pulmonary disease, pulmonary fibrosis, pulmonary infection in the last 3 months, or history of aspiration,
7. History of unexplained jaundice by subject report,
8. History of Hepatitis A, B, or C or HIV by subject report,
9. History of stem cell therapy,
10. History of immune modulator therapy (e.g., corticosteroids, IV immunoglobulin, immunosuppressive chemotherapeutic agents, plasma exchange, GM-CSF, MCSF, interferons, infliximab, natalizumab, fingolimod [GILENYA], masitinib, ibudilast, tofacitinib citrate [XELJANZ], or any other approved drugs intended to affect the immune system) within 12 weeks of Screening Visit. Locally-acting corticosteroids (inhaled, intranasal, and topical) are permitted,
11. Participation in an experimental drug trial (of agents other than immune modulators) within 12 weeks prior to Screening Visit. Observational trials with no intervention are acceptable provided permission from the other study sponsor is obtained in writing,
12. Systolic blood pressure < 100 mm Hg or > 160 mm Hg, diastolic blood pressure > 98 mm Hg. Patients on stable treatment for at least 3 months for hypertension are allowed as long as they meet entry criteria,
13. Hematocrit < 33%, platelet count < lower limit of normal, or neutrophil count < 1,500/mm3,
14. Estimated creatinine clearance (eCCr) < 50 mL/minute by Cockcroft-Gault Formula,
15. Elevated aspartate aminotransferase (AST) or alanine aminotransferance (ALT) greater than 3 times the upper limit of normal,
16. Pregnant or lactating females,
17. Have any condition which, in the opinion of the investigator, would put the subject at risk by participating in this study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Inflammatory monocyte-associated biomarkers | 7 days
  The primary endpoint is changes from baseline at 1 and 7 days following dosing in percent monocyte expression levels of CD16 and HLA-DR.

SECONDARY OUTCOMES:
Adverse Events | 7 days
  The secondary endpoint is reported and observed adverse events following dosing and at 1 and 7 days post-infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Beau Nakamoto, MD PhD, Principal Investigator — University of Hawaii
Locations (1):
- University of Hawaii Clinics at Kakaako, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

REFERENCES:
- [Background] Miller RG, Block G, Katz JS, Barohn RJ, Gopalakrishnan V, Cudkowicz M, Zhang JR, McGrath MS, Ludington E, Appel SH, Azhir A; Phase 2 Trial NP001 Investigators. Randomized phase 2 trial of NP001-a novel immune regulator: Safety and early efficacy in ALS. Neurol Neuroimmunol Neuroinflamm. 2015 Apr 9;2(3):e100. doi: 10.1212/NXI.0000000000000100. eCollection 2015 Jun. PMID 25884010
- [Background] Miller RG, Zhang R, Block G, Katz J, Barohn R, Kasarskis E, Forshew D, Gopalakrishnan V, McGrath MS. NP001 regulation of macrophage activation markers in ALS: a phase I clinical and biomarker study. Amyotroph Lateral Scler Frontotemporal Degener. 2014 Dec;15(7-8):601-9. doi: 10.3109/21678421.2014.951940. Epub 2014 Sep 5. PMID 25192333
- [Background] Zhang R, Miller RG, Madison C, Jin X, Honrada R, Harris W, Katz J, Forshew DA, McGrath MS. Systemic immune system alterations in early stages of Alzheimer's disease. J Neuroimmunol. 2013 Mar 15;256(1-2):38-42. doi: 10.1016/j.jneuroim.2013.01.002. Epub 2013 Feb 4. PMID 23380586
- [Background] Pey P, Pearce RK, Kalaitzakis ME, Griffin WS, Gentleman SM. Phenotypic profile of alternative activation marker CD163 is different in Alzheimer's and Parkinson's disease. Acta Neuropathol Commun. 2014 Feb 14;2:21. doi: 10.1186/2051-5960-2-21. PMID 24528486